CLINICAL TRIAL: NCT00688662
Title: A Phase III Randomized Multicenter Clinical Trial of Sphincterotomy for the Treatment of SOD III Patients
Brief Title: Evaluating Predictors & Interventions in Sphincter of Oddi Dysfunction
Acronym: EPISOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Peter Cotton, Study Chair, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK074739; U01DK074739 (NIH)
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Sphincter of Oddi Dysfunction
Keywords: Sphincter of Oddi Dysfunction; Pancreatitis; Sphincterotomy
MeSH Terms: conditions — Sphincter of Oddi Dysfunction; Pancreatitis | interventions — Cholangiopancreatography, Endoscopic Retrograde; Sphincterotomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.ERCP with sphincterotomy (Active Comparator): ERCP with sphincterotomy: cutting the biliary sphincter muscle (sphincterotomy)
  Interventions: Procedure: ERCP with sphincterotomy
- 2.ERCP without sphincterotomy (Placebo Comparator): ERCP without cutting the biliary sphincter muscle (sphincterotomy)
  Interventions: Procedure: ERCP without sphincterotomy

INTERVENTIONS:
Procedure: ERCP with sphincterotomy — cutting the biliary sphincter muscle (sphincterotomy)
  Arms: 1.ERCP with sphincterotomy
Procedure: ERCP without sphincterotomy — ERCP with sphincter manometry, but no sphincterotomy
  Arms: 2.ERCP without sphincterotomy

SUMMARY:
The Evaluating Predictors & Interventions in Sphincter of Oddi Dysfunction(SOD) study (EPISOD) is a randomized sham-controlled study of biliary and pancreatic sphincterotomy as treatment for patients with pain after cholecystectomy fitting the criteria for sphincter of Oddi dysfunction type III.

DETAILED DESCRIPTION:
Clinical Trial Phase: Phase III

Study Sites Seven clinical centers in US

Study Period Planned enrollment period - 3 years

Planned duration of the study - 5 years

Study Population SOD III Patients

Primary Study Objective: To ascertain whether subjects with SOD III respond to sphincterotomy,

Secondary Study Objectives

To evaluate:

* the association between the results of Sphincter of Oddi Manometry (SOM) (abnormal/normal) and the primary outcome (success/failure);
* the success rate (as defined in the primary) of subjects who receive biliary sphincterotomy alone versus subjects who receive both biliary and pancreatic sphincterotomy in the subgroup of patients with manometrically proven hypertension of the pancreatic sphincter;
* the effects of pre-specified prognostic factors on the primary outcome;
* anxiety and depression scores over time and their relation to study outcomes;
* the economic impact of SOD III, and of endoscopic sphincterotomy in patients with SOD III; and, to,
* conduct a careful follow-up study (EPISOD2) of standard of care treatment (separate protocol).

Study Design The EPISOD Trial is a parallel, randomized, double-blinded, sham-controlled, multicenter Phase III clinical trial of endoscopic sphincterotomy as treatment for adults 18 to 65 years of age diagnosed with SOD III.

Sample Size A minimum of 214 subjects will be randomized using a 2:1 allocation in favor of sphincterotomy and will be followed for 12 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with the clinical syndrome of SOD, as defined by the Modified Functional Biliary Disorders Module of the Rome III criteria
2. Pain burden of Grade 3 or higher on RAPID Questionnaire.
3. Cholecystectomy more than 90 days before enrollment.
4. Laboratory Tests: Results of blood tests taken within 1 week preceding the baseline visit and any others available from the preceding 6 months (post-cholecystectomy):Direct bilirubin, alkaline phosphatase, amylase and lipase results must be no greater than 2 X the upper level of normal.Transaminase levels can be no more than 3 X upper limit of normal. If the transaminases are elevated (<2X ULN) in association with a pain attack, they cannot have returned to normal within 3 days.
5. Normal abdominal imaging by CT or MR/MRCP with bile duct reported at ≤9mm.
6. Upper endoscopy examination without findings to explain the pain.
7. Pain persisting despite a one trial of acid suppressant medications for one month (if tolerated).
8. Pain persisting despite a trial of antispasmodics.
9. Subjects on antidepressants for pain control (not required) should be taking them for a minimum of one month prior to the baseline assessment.

9.Patients with SOD with depressive and/or anxiety disorders who receive psychopharmacologic treatment must be on stable medication dose for at least 6 weeks.

10.Access to a telephone. 11.Must be able to speak, read, and write English. 12.Signed and dated informed consent.

Exclusion Criteria:

1. Prior ERCP treatment.
2. Age < 18 or Age > 65.
3. Pregnancy: Women who are pregnant at the time of Screening* will be excluded from the study. (*Note: Women who become pregnant AFTER the Baseline Visit/ERCP will be allowed to remain in the study for telephone follow-up visits).
4. Prior gastric resection or surgery involving biliary diversion.
5. Prior diagnosis of acute pancreatitis (lipase >3 x ULN) including post-ERCP pancreatitis, or of chronic pancreatitis by radiological imaging, EUS 5 or more criteria, or Cambridge criteria moderate or more on ERCP.
6. Daily use of prescription analgesics over the previous month.
7. Abdominal discomfort every day for the past month at level of 3 or more on a scale of 1-10.
8. Presence of significant psychiatric disorders:

   1. Lifetime psychotic disorders, bipolar disorder;
   2. Substance use disorders within 6 months;
   3. Eating disorders within 2 years
   4. Moderate & severe depression defined by BDI-II (Beck Depression Inventory) cutoff scores >22 (unless receiving stable psychiatric therapy for six weeks); and/or,
   5. Suicidal risk (equal to or greater than "low") using MINI suicide section or a score of greater than 0 on question 9 of the BDI.
9. The total number of days in the previous 3 months that the subject has taken prescription analgesics due to episodes of abdominal pain is greater than the total number of days the subject had episodes of abdominal pain.
10. Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation.

ERCP Criteria:

1. Pancreas divisum (complete or partial) (known or discovered at study ERCP).
2. Any pathology found at ERCP (except sphincter hypertension).
3. Failed pancreatic manometry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2008-07; Primary Completion 2013-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Romagnuolo, MD, Principal Investigator — Medical Universtiy of South Carolina; Martin Freeman, MD, Principal Investigator — University of Minnesota; Richard Kozarek, MD, Principal Investigator — Virginia Mason Medical Center; Evan Fogel, MD, Principal Investigator — Indiana University; Peter Cotton, MD, Study Chair — MUSC Digestive Disease Center; Paul Tarnasky, MD, Principal Investigator — Digestive Health Associates of Texas; Giuseppe Aliperti, MD, Principal Investigator — Midwest Therapeutic Endoscopy Consultants; Priya Jamidar, MD, Principal Investigator — Yale University; Jose Serrano, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (7):
- United States (7):
  - Yale University, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Midwest Therapeutic Endoscopy Consultants, St Louis, Missouri
  - Medical University of South Carolina Digestive Disease Center, Charleston, South Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Yaghoobi M, Pauls Q, Durkalski V, Romagnuolo J, Fogel EL, Tarnasky PR, Aliperti G, Freeman ML, Kozarek RA, Jamidar PA, Wilcox CM, Elta GH, Hawes RH, Wood-Williams A, Cotton PB. Incidence and predictors of post-ERCP pancreatitis in patients with suspected sphincter of Oddi dysfunction undergoing biliary or dual sphincterotomy: results from the EPISOD prospective multicenter randomized sham-controlled study. Endoscopy. 2015 Oct;47(10):884-90. doi: 10.1055/s-0034-1392418. Epub 2015 Jul 10. PMID 26165739
- [Derived] Cotton PB, Durkalski V, Romagnuolo J, Pauls Q, Fogel E, Tarnasky P, Aliperti G, Freeman M, Kozarek R, Jamidar P, Wilcox M, Serrano J, Brawman-Mintzer O, Elta G, Mauldin P, Thornhill A, Hawes R, Wood-Williams A, Orrell K, Drossman D, Robuck P. Effect of endoscopic sphincterotomy for suspected sphincter of Oddi dysfunction on pain-related disability following cholecystectomy: the EPISOD randomized clinical trial. JAMA. 2014 May;311(20):2101-9. doi: 10.1001/jama.2014.5220. PMID 24867013
- [Derived] Romagnuolo J, Cotton PB, Durkalski V, Pauls Q, Brawman-Mintzer O, Drossman DA, Mauldin P, Orrell K, Williams AW, Fogel EL, Tarnasky PR, Aliperti G, Freeman ML, Kozarek RA, Jamidar PA, Wilcox CM, Serrano J, Elta GH. Can patient and pain characteristics predict manometric sphincter of Oddi dysfunction in patients with clinically suspected sphincter of Oddi dysfunction? Gastrointest Endosc. 2014 May;79(5):765-72. doi: 10.1016/j.gie.2013.11.037. Epub 2014 Jan 25. PMID 24472759
- [Derived] Cotton PB, Durkalski V, Orrell KB, Brawman-Mintzer O, Drossman DA, Wilcox CM, Mauldin PD, Elta GH, Tarnasky PR, Fogel EL, Jagganath SB, Kozarek RA, Freeman ML, Romagnuolo J, Robuck PR. Challenges in planning and initiating a randomized clinical study of sphincter of Oddi dysfunction. Gastrointest Endosc. 2010 Nov;72(5):986-91. doi: 10.1016/j.gie.2010.08.022. PMID 21034899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from medical clinics in 6 gastroenterology referral centers in USA between August 6 2008 and March 23 2012.
Groups:
- 1.ERCP With Sphincterotomy: Endoscopic Retrograde CholangioPancreatography (ERCP) with biliary and/or pancreatic sphincterotomy
- 2. ERCP Without Sphincterotomy:: Endoscopic Retrograde CholangioPancreatography (ERCP) without biliary and/or pancreatic sphincterotomy
Period: Overall Study
Arm/Group | 1.ERCP With Sphincterotomy | 2. ERCP Without Sphincterotomy:
Started | 141 | 73
Completed | 118 | 55
Not Completed | 23 | 18

BASELINE CHARACTERISTICS:
Groups:
- 1. ERCP With Sphincterotomy: Endoscopic Retrograde CholangioPancreatography (ERCP) with sphincter manometry and biliary and/or pancreatic sphincterotomy and pancreatic stenting
- 2. ERCP Without Sphincterotomy: Endoscopic Retrograde CholangioPancreatography(ERCP) with sphincter manometry and pancreatic stenting, but without sphincterotomy
- Total: Total of all reporting groups
Arm/Group | 1. ERCP With Sphincterotomy | 2. ERCP Without Sphincterotomy | Total
Number analyzed (Participants) | 141 | 73 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 141 | 73 | 214
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 69 | 197
  Male | 13 | 4 | 17
Region of Enrollment [Number; unit: participants]
  United States | 141 | 73 | 214

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Success
Description: The primary outcome was a dichotomous (success/failure) variable. Success was defined as patients having a RAPID score of <6 days at months 9 and 12 post-procedure, without re-intervention and without use of prescription analgesics during months 10, 11 and 12 unless used for non-abdominal pain for no more than 14 days. The subject was considered a failure if the 12-month RAPID score was missing or collected outside the acceptable window. If the 9-month RAPID was missing, or outside of the window, then the 6-month value was used when available.
Time Frame: 1 year
Population: The primary analysis was conducted with the intention-to-treat population defined as all randomized patients.
Measure: Number (95% Confidence Interval); unit: percentage of paricipants with success
Groups:
- 2. ERCP Without Sphincterotomy: ERCP without sphincterotomy: ERCP with sphincter manometry, but no sphincterotomy
Arm/Group | 1.ERCP With Sphincterotomy | 2. ERCP Without Sphincterotomy
Number analyzed (Participants) | 141 | 73
percentage of paricipants with success | 23 [15.8 to 29.6] | 37 [25.9 to 48.1]
Statistical Analysis 1: Comparison: 1.ERCP With Sphincterotomy vs 2. ERCP Without Sphincterotomy; The trial was designed to test for an overall absolute difference of at least 30% in the primary outcome ('success') in patients treated with sphincterotomy compared to those treated with sham. Using a 2:1 allocation, an assumed 10% non-adherence rate, and one interim analysis for efficacy using O'Brien and Fleming boundaries and futility using conditional power, the study required 214 patients to be randomized to ensure greater than 90% likelihood of identifying this difference; Test type: Superiority or Other; p = 0.01, Regression, Logistic — The primary analysis was conducted using a logistic regression model with treatment group as the factor of interest and clinical center and PSH status as covariates. A Wald test using a two-tailed significance level of 0.0499 was conducted; Adjusted and unadjusted risk differences with two-sided 95% confidence intervals are reported in the manuscript; Risk Difference (RD) = -15.6, 95% CI 2-sided [-28.0 to -3.3] — The unadjusted risk difference and confidence interval was -14.3% (-27.3%, -1.2%)

2. Secondary Outcome: Percentage of Patients With a Successful Primary Outcome, Out of Those With Abnormal Sphincter Manometry.
Description: Successful outcome was defined using the primary outcome definition of success at 12 months post randomization. Abnormal sphincter manometry was determined as a basal pressure of more than 40mm Hg in both leads.
Time Frame: 1 year
Population: Participants with abnormal sphincter manometry
Measure: Number; unit: percentage of participants with success
Arm/Group | 1.ERCP With Sphincterotomy | 2.ERCP Without Sphincterotomy
Number analyzed (Participants) | 110 | 52
percentage of participants with success | 24 | 33
Statistical Analysis 1: Comparison: 1.ERCP With Sphincterotomy vs 2.ERCP Without Sphincterotomy; Only patients with abnormal manometry were included in this subgroup analysis; Test type: Superiority or Other; A confidence interval approach was used for examining this outcome; Risk Difference (RD) = -9, 95% CI 2-sided [-24.1 to 5.9]

ADVERSE EVENTS:
Time Frame: One year after randomization
Arm/Group | 1.ERCP With Sphincterotomy | 2. ERCP Without Sphincterotomy
Serious Adverse Events (participants affected / at risk) | 16/141 | 12/73
Other Adverse Events (participants affected / at risk) | 0/141 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1.ERCP With Sphincterotomy (N=141) | 2. ERCP Without Sphincterotomy (N=73)
Pancreatitis (Gastrointestinal disorders) | 15 | 11
Perforation (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No